CLINICAL TRIAL: NCT04804878
Title: Morehouse Total Cancer Care Protocol: A Lifetime Partnership With Patients Who Have or May be at Risk of Having Cancer
Brief Title: Morehouse Total Cancer Care Protocol
Acronym: MSMTCC
Status: Recruiting | Type: Observational
Sponsor: Morehouse School of Medicine (Other)
Responsible Party: Principal Investigator, James Lillard, PhD, Professor of Microbiology, Biochemistry, & Immunology, Morehouse School of Medicine
Other Study IDs: 841718
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Cancer; Cancer Risk
MeSH Terms: conditions — Neoplasms | interventions — Histocompatibility Testing; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Biospecimens collected under TCC protocol can include excess tissue, fluid or blood removed during a clinical procedure, tissue collected as part of clinical care, and research specific collection. Other biological samples, such as saliva, sputum, urine, feces, hair, surface skin swabs, etc., may be collected as part of the TCCP if the collection meets criteria for minimal risk and/or is part of the patient's routine standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biospeciman Repository and Data Collection: Patients with cancer or who are at risk of having cancer who have given consent to have blood, tissue, other biological samples and their associated data (survey data, medical records data, cancer registry data, and other related data) collected and stored for the advancement of medicine.
  Interventions: Procedure: Collection of blood, tissue, and other biological samples.; Other: Medical Chart Review

INTERVENTIONS:
Procedure: Collection of blood, tissue, and other biological samples. — Behavioral health assessments, including quality of life.
  Other Names: Surveys
Other: Medical Chart Review — Health data abstracted directly from patient's health records

SUMMARY:
The overall objective of the Morehouse Total Cancer Care study is to develop an improved standard of cancer care by facilitating new biomarker and drug target discovery, informatics solutions, clinical trials, and "personalized medicine" for our community oncology partners (i.e., community hospital systems, and other cancer care providers). To bring new translational research to the community, Morehouse School of Medicine has initiated the Total Cancer Care Program (TCCP). The TCCP establishes a unique collection of blood, tissue, other biological samples and their associated data (survey data, medical records data, cancer registry data, and other related data) from thousands of African American cancer patients, survivors, or those at risk of having cancer. This is not a treatment trial, but a longitudinal study designed to create a centralized cancer biorepository for precision medicine.

DETAILED DESCRIPTION:
Through this protocol, Morehouse School of Medicine and its partners will establish and maintain a unique repository of blood, tissue, other biological samples and their associated data (survey data, medical records data, cancer registry data, and other related data) collected from thousands of patients 18 years of age or older who have cancer or are at risk of developing cancer. In this protocol, investigators require an informed consent of patients to study their answers to survey questions that may be collected as part of their regular clinical care, permission to study their medical and related records, and permission to collect excess tissues removed at the time of planned surgery, an additional tumor sampling (needle passes) at the time of planned diagnostic biopsies, previously collected, stored tumor tissue (if available), blood, and/or other biological samples. Additional research tumor samples may be collected at the time of any diagnostic needle biopsy or endoscopic biopsy or, if available, patient tissue from a previous procedure will be obtained and utilized as needed. Clinical and related data will be collected on all patients from the time of initial entry into the study and will continue for life.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older.
2. Diagnosed with cancer, or at risk for cancer. This includes anyone in the general population, but our primary focus will be on patients with a cancer diagnosis.
3. Able to understand and sign the TCCP Informed Consent and Research Authorization form directly or through an authorized representative. The Informed Consent and Research Authorization will be available in both English and Spanish languages

Exclusion Criteria:

None

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who have cancer or are at risk of developing cancer.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2035-04 (Estimated); Study Completion 2037-04 (Estimated)

PRIMARY OUTCOMES:
Improve Standard of Cancer Care | Time Frame: up to 20 years
  Establish a longitudinal clinical and related data and tissue repository that will contain cancer predisposing risk factors via surveys and questionnaires.
Improve Standard of Cancer Care | Time Frame: up to 20 years
  Establish a longitudinal clinical and related data repository that will contain quality of life care via surveys and questionnaires
Improve Standard of Cancer Care | Time Frame: up to 20 years
  Establish a longitudinal tissue repository that will contain blood, tissue, and other biological samples other biological samples and associated clinical data collected from consenting patients.

CONTACTS AND LOCATIONS:
Overall Officials: James W Lillard, PhD, Principal Investigator — Morehouse School of Medicine
Locations (1):
- Morehouse School of Medicine, Atlanta, Georgia, United States